CLINICAL TRIAL: NCT07187622
Title: The Effect of Education Given to Mothers to Prevent Neonatal Jaundice on the Knowledge Level and Frequency of Jaundice Development
Brief Title: The Effect of Neonatal Jaundice Education on Mothers' Knowledge Level and the Incidence of Jaundice Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Gülzade Uysal, Associate Professor, PhD, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/08-16
Record Dates: First submitted 2025-07-14; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Education
Keywords: Knowledge level; Pregnant women; Newborn; Neonatal jaundice; Education
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Intervention Model Description: research and control group
Masking Description: research and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- research group (Experimental): After the first application of the scale, mothers in the research group will be given education about neonatal jaundice using a direct instruction method with an education booklet in line with the "Education content plan". The newborn jaundice status of the babies will be examined.
  Interventions: Other: examine the impact of education
- control group (No Intervention): Mothers in the control group will not be given education.

INTERVENTIONS:
Other: examine the impact of education — The mothers in the study group were given education about neonatal jaundice and were trained to increase the mothers' knowledge level and to prevent neonatal jaundice.
  Arms: research group

SUMMARY:
This study was a randomised controlled trial conducted to determine the effect of the training given to mothers who gave birth by caesarean section in the obstetrics and gynaecology service clinic of Sultanbeyli State Hospital on the level of knowledge and the frequency of jaundice development. All participants who fulfil the inclusion criteria (86 in total) will be included in the study. The 'maternal data collection form' and 'information form on neonatal jaundice' will be applied to the pregnant women as a pre-test. Training will be planned for the participants in the intervention group in 2 sessions. Mothers in the control group will not receive this planned training. On the day of discharge, the 'neonatal jaundice information form' will be filled in again by the participants and the information scores will be recorded. After the intervention group is discharged, they will be called by telephone and jaundice symptoms will be questioned. After 1 month, the 'information form on neonatal jaundice' and 'neonatal follow-up form' will be filled in both groups and the information will be recorded.

DETAILED DESCRIPTION:
Jaundice, or hyperbilirubinemia, is a condition in which the sclera, skin and mucous membranes appear yellow with an increase in bilirubin level in the blood. Neonatal jaundice is one of the main reasons for hospitalisation and it is still an important health problem in Turkey. In a study, it was reported that 6.4% of hospitalised infants had severe hyperbilirubinemia.

Neonatal jaundice is observed in 80% of preterm babies and 60% of term babies. Jaundice becomes visible when the total bilirubin level is above 5 mg/dl. Jaundice is visible in 60% of newborns born on time. The course of the disease is mild, disappears spontaneously in the third week in preterm newborns and in the second week in term newborns without the need for any treatment.

Although neonatal jaundice is generally seen as a temporary and harmless condition, it can seriously harm the baby's health when left untreated. When high bilirubin levels are not intervened, serious neurological damage occurs. In order to prevent possible damage, close monitoring of the newborn is of great importance for early diagnosis and treatment of neonatal jaundice. Neonatal jaundice usually reaches its peak on the 5th and 7th days of the baby. While most term babies without any problems are discharged before these time periods, most neonatal jaundice is seen at home. Mothers who care for discharged babies are the first to observe jaundice. When each newborn is discharged, appropriate follow-up for jaundice should be performed considering the risk factors for hyperbilirubinemia, and families should be given information and written guidelines about jaundice.

It is possible to prevent neonatal jaundice by early diagnosis and application of appropriate intervention methods. In this direction, it is of great importance that mothers have sufficient knowledge about jaundice. Early recognition of jaundice symptoms by mothers reduces the risk of serious complications that may develop in the newborn by enabling them to apply to healthcare institutions without delay. However, scientific studies have revealed that the majority of mothers have a widespread lack of knowledge about neonatal jaundice. Implementation of planned and comprehensive training programmes for mothers by healthcare professionals stands out as an effective strategy in the fight against neonatal jaundice. Such trainings improve the knowledge level of mothers, enabling them to recognise the symptoms of jaundice in a timely manner and take necessary precautions.

Methods:

The study will be examined with a randomized controlled design to determine the effect of the education given to mothers who gave birth by cesarean section at the gynecology and obstetrics clinic of Sultanbeyli State Hospital on the level of knowledge and the frequency of jaundice development.

The study will be randomly selected by lottery after obtaining the necessary permissions.

The universe of the study will be conducted between November 2023 and November 2024 at the gynecology and obstetrics department of Istanbul Sultanbeyli State Hospital.

The sample calculation of the study was made with the G-power 3.1 package program. For this purpose, the data in the study of Bekmezci (2023), which is a similar study, were taken into account and the effect size and sample calculation were made. In the sample calculation, it was determined that a total of 78 participants, 39 in each group, were included with a margin of error of .05, a confidence interval of .95 and an effect size of .38. Considering that there may be a loss from the sample during the study period, the sample size was increased by 10% and a total of 86 participants (Intervention: 43, Control: 43) were included in the study. A simple randomization system was used for selection in the study.

Data Collection Tools 'Informed Consent Form', "Maternal data collection form" including the information of the mother, "Information form on neonatal jaundice" to determine the knowledge level of the mothers, "Neonatal follow-up form" including the information of the baby, and "Training booklet on neonatal jaundice" presenting the content of the training subjects were used.

Informed Consent Form It is a form in which the mothers participating in the research accept the research, the contact information of the researcher and information about the research is included.

Mother Data Collection Form The form consists of 10 questions including information about the sociodemographic status, employment status, education level, blood group, family type of the mothers in line with the literature and there is also a table in which the knowledge score of the mothers about jaundice will be recorded.

Information Form on Neonatal Jaundice The form was designed to measure mothers' level of knowledge about neonatal jaundice. Questions about neonatal jaundice were developed by using the literature. It was formed as a form consisting of a total of 30 true-false questions including questions about the definition of neonatal jaundice, how common it is, when it occurs, risk factors, symptoms and signs, causes, diagnosis and treatment, things to be considered in neonatal jaundice, how mothers can protect their babies from neonatal jaundice, wrong traditional methods applied in neonatal jaundice. The calculation was made by giving '1' point for each correct answer and '0' point for each wrong answer. The scoring is prepared in such a way that a minimum of 0 and a maximum of 30 points are obtained.

Newborn Monitoring Form The form consisted of 11 questions to be asked to both the study and control groups, including questions about the descriptive information of the infant and jaundice status, which were formed in line with the literature. In order to ensure that the jaundice symptoms and findings of the babies in the intervention group were closely monitored by the mothers, they were called by telephone on the 3rd, 5th, 7th, 10th and 15th days and the table containing the jaundice symptoms and findings consisting of 8 questions was included in this form.

Training Booklet on Neonatal Jaundice In the training booklet, a training booklet was prepared under the titles of what is neonatal jaundice, how common it is, when it occurs, what are the risk factors, what are the symptoms, how can we understand neonatal jaundice, how can you protect your baby from neonatal jaundice, what is the diagnosis and treatment, and this booklet was planned to be given to families. The content of the booklet was created in line with expert opinions and used Application The mothers participating in the study were included in 2 groups as intervention and control groups. After the hospitalisation procedures of the pregnant woman who applied to the service were completed, information about the service was given and the pregnant woman was taken to her room. After the necessary treatment and information were given to the pregnant woman who was hospitalised, information about the study was given and 'Informed Consent Form' was taken from the pregnant women who wanted to participate in the study and informed about the process. Pregnant women who accepted the study were asked to fill out the 'Maternal Data Collection Form' as a pre-test and the 'Information Form on Neonatal Jaundice' to measure the level of knowledge of mothers about jaundice of the newborn. Preoperative preparation of the pregnant woman was done and she was taken to the operating theatre for caesarean section. Breastfeeding training, which is in the service routine, was given to the mother coming from caesarean section by the lactation nurse and the mother was supported by initiating the first breastfeeding. The 'Newborn follow-up form' containing the baby's information is completed.

Intervention Group Practice

* With the stabilisation of the mother's condition, on the first day of hospitalisation, the mother was interviewed one-to-one in her own room, and training was given on what neonatal jaundice is, how common it is, when jaundice occurs, and what are the risk factors for jaundice as the first session of the training. The training lasted 30 minutes on average. 'Education Booklet on Jaundice of the Newborn' was given to the mother.
* On the second day of hospitalisation, the training given to the mother on the first day in her room was repeated in general and the training including the signs and symptoms of jaundice, how to understand jaundice, how to protect our baby from jaundice, diagnosis and treatment of neonatal jaundice was given in an average of 60 minutes and the questions asked by the mother were answered.
* How to control the skin of the baby was explained practically and after discharge, she was asked to visually monitor the baby's skin in terms of jaundice every day on a white sheet, naked in daylight.
* The training consisted of 2 sessions. Then, the 'Information Form on Neonatal Jaundice' was repeated on the day of discharge for all mothers who received the training and the mother was discharged. These mothers were also given discharge training as part of the ward routine.
* Mothers who received at least 2 sessions of planned neonatal jaundice training were given an appointment 1 month later for the application of the post-test.
* Mothers who were discharged after receiving neonatal jaundice training were called by phone on the 3rd, 5th, 7th, 10th, 15th day of the baby and information about the jaundice status of the baby was obtained, and the 8 signs and symptoms of neonatal jaundice in the 'Neonatal Follow-up Form' were filled in +/- in line with the information provided by the mothers. Mothers who encountered problems were referred to the paediatrician and the lactation polyclinic of the hospital.
* Mothers were invited to the institution 1 month after the training. In order to measure the knowledge score of the mothers, the 'Information Form on Neonatal Jaundice' was repeated to the mothers in the baby room as a post-test. The scores of the mothers were recorded on the follow-up form. The neonatal jaundice status of the babies was recorded in the 'Neonatal Follow-up Form'. In case the baby was hospitalised in the neonatal intensive care unit due to jaundice, the number of hospitalisation days and hospitalisation bilirubin level parameters included in the questions were recorded in the 'Neonatal follow-up form' by looking at the hospital's HIS module.
* The training booklet remained with the mothers during and after the training. Control Group Practice
* The 'Information Form on Neonatal Jaundice' was repeated on the day of discharge for the mothers who accepted the study during hospitalisation but were not given planned neonatal jaundice education. These mothers were only given discharge and breastfeeding education, which were in the ward routine.
* On the day of discharge, an appointment was arranged for 1 month later for the administration of the post-test.
* One month after discharge, the mothers who made an appointment for the hospital visit were taken to the baby's room and the 'Information Form on Neonatal Jaundice' and the part of the 'Neonatal Follow-up Form' containing information about the baby, which included questions about the jaundice status of the baby, were filled in for the post-test. In case the baby was hospitalised in the neonatal intensive care unit due to jaundice, the number of days of hospitalisation and hospitalisation bilirubin level parameters included in the questions were recorded in the 'Neonatal follow-up form' by looking at the hospital's HIS module.
* The scores of the mothers who completed the information form 1 month after discharge were recorded in the follow-up form.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who gave birth by planned cesarean section,
* Mothers who did not receive planned training on neonatal jaundice,
* Having been hospitalized for at least 2 days and having attended training at least 2 times until the day of discharge,
* Being willing and willing to participate in the study,
* Mothers who have the ability to read, write and understand Turkish,
* Not having a psychological or mental disability

Exclusion Criteria:

* Mothers who did not attend the training or were discharged before 2 days,
* Mothers who were admitted to the ward with an emergency cesarean section,
* Having a risky pregnancy,
* The baby being admitted to the intensive care unit during the hospitalization period (within 48 hours),
* The baby being admitted to the intensive care unit with a diagnosis other than neonatal jaundice after discharge,
* Not being able to contact during the training process,
* Mothers who did not attend the final test 1 month after the training

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in neonatal jaundice knowledge scores of the trained group after the training | Measurements will be made before the training, at discharge and 1 month after the training
  After the planned 2-day training, the mothers' knowledge level about neonatal jaundice was determined with the "Neonatal jaundice knowledge form". The increase in the knowledge score indicates that the mothers' knowledge level about jaundice increased. The total score range of the 30-item scale varies between 0 and 30. The lowest score that can be obtained from the scale is "0" and the highest score is "30".

SECONDARY OUTCOMES:
Change in jaundice status of newborns after the education | 1 month after education
  After the 2-day education, mothers will be called on the 3rd, 5th, 7th, 10th and 15th days of discharge and asked about jaundice symptoms and findings consisting of 8 questions. After 1 month, the "Neonatal Follow-up Form" will be filled.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia MENGÜTAY, Principal Investigator — Okan University School of Nursing İstanbul, Turkey
Locations (1):
- Okan University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Plan to Share IPD:

REFERENCES:
- [Background] Rathore S, Kumar Vk C, R S. A critical review on neonatal hyperbilirubinemia-an Ayurvedic perspective. J Ayurveda Integr Med. 2020 Apr-Jun;11(2):190-196. doi: 10.1016/j.jaim.2018.08.006. Epub 2019 Oct 15. PMID 31628007
- [Background] Erdeve O, Okulu E, Olukman O, Ulubas D, Buyukkale G, Narter F, Tunc G, Atasay B, Gultekin ND, Arsan S, Koc E; Turkish Neonatal Jaundice Registry Collabolators. The Turkish Neonatal Jaundice Online Registry: A national root cause analysis. PLoS One. 2018 Feb 23;13(2):e0193108. doi: 10.1371/journal.pone.0193108. eCollection 2018. PMID 29474382
- [Background] Anderson NB, Calkins KL. Neonatal Indirect Hyperbilirubinemia. Neoreviews. 2020 Nov;21(11):e749-e760. doi: 10.1542/neo.21-11-e749. PMID 33139512
- [Background] Maisels MJ, Watchko JF. Improving post-discharge neonatal surveillance for the jaundiced newborn. Acta Paediatr. 2020 May;109(5):872-873. doi: 10.1111/apa.15154. Epub 2020 Feb 3. No abstract available. PMID 32017238
- [Background] Huang Y, Chen L, Wang X, Zhao C, Guo Z, Li J, Yang F, Cai W. Maternal knowledge, attitudes and practices related to neonatal jaundice and associated factors in Shenzhen, China: a facility-based cross-sectional study. BMJ Open. 2022 Aug 24;12(8):e057981. doi: 10.1136/bmjopen-2021-057981. PMID 36002214
- [Background] Wennberg RP, Oguche S, Imam Z, Farouk ZL, Abdulkadir I, Sampson PD, Slusher TM, Bode-Thomas F, Toma BO, Yilgwan CS, Shwe D, Ofakunrin AO, Diala UM, Isichei C, Pam V, Hassan Z, Abdullahi SU, Usman F, Jibir BW, Mohammed IY, Usman HA, Abdusalam M, Kuliya-Gwarzo A, Tsiga-Ahmad FI, Umar L, Ogala WN, Abdullahi F, Hassan L, Purdue S, Lund T, Coda-Zabetta CD. Maternal Instruction About Jaundice and the Incidence of Acute Bilirubin Encephalopathy in Nigeria. J Pediatr. 2020 Jun;221:47-54.e4. doi: 10.1016/j.jpeds.2020.01.050. Epub 2020 Mar 4. PMID 32145967
- [Background] Amegan-Aho KH, Segbefia CI, Glover NDO, Ansa GA, Afaa TJ. Neonatal Jaundice: awareness, perception and preventive practices in expectant mothers. Ghana Med J. 2019 Dec;53(4):267-272. doi: 10.4314/gmj.v53i4.3. PMID 32116337
- [Background] Alinaitwe B, Francis N, Ngabirano TD, Kato C, Nakamya P, Uwimbabazi R, Kaplan A, McCoy M, Ayebare E, Winter J. Delivery of a post-natal neonatal jaundice education intervention improves knowledge among mothers at Jinja Regional Referral Hospital in Uganda. PLoS One. 2024 Apr 4;19(4):e0301512. doi: 10.1371/journal.pone.0301512. eCollection 2024. PMID 38574088